CLINICAL TRIAL: NCT01923519
Title: Study of Genic Expression Profiles of the Epithelium of the Nose and Bronchi in Healthy and Allergic Subjects
Acronym: GENEBRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 13-PP-06
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-07

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- allergic rhinitis (Experimental)
  Interventions: Procedure: bronchofiberscopy
- allergic rhinitis and asthma (Experimental)
  Interventions: Procedure: bronchofiberscopy
- witnesses (Experimental)
  Interventions: Procedure: bronchofiberscopy

INTERVENTIONS:
Procedure: bronchofiberscopy

SUMMARY:
The respiratory epithelium plays a leading role in the development of allergic respiratory disease with barrier function alteration, its repair mechanisms, of anti-viral fight and the ability to induce by itself Th2 responses. The majority of allergic asthmatic patients have reached concomitant ENT: the concept of "one airway, one disease." Access to this material of epithelial study in the different phenotypes of the disease appears to be crucial. Nasal and bronchial epithelial tissues reveal essential differences in particular related to their environment (remodeling less intense and a lower sensitivity to the virus in the nose), but they nevertheless share many common cellular characteristics.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years and <30 years
* isolated allergic rhinitis according to clinical criteria ARIA
* absence of asthma whose diagnosis is made based on clinical criteria or mild to moderate persistent asthma controlled with a diagnosis is made based on clinical criteria

Exclusion Criteria:

* recent rhino-bronchial infection (<6 weeks)
* asthma exacerbation in the previous 6 weeks
* Chronic disease may in the opinion of the investigators interfere with the results of the study or expose them to additional risk.
* Treatment with nasal corticosteroids, inhaled or systemic in the past 6 weeks
* Current smoking no history of smoking or not smoking for at least 12 months and weaned smoking history <5 pack-years)
* Special Needs

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
genic expression profile of the epithelium | 3 months after inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Pasteur, Nice, France

REFERENCES:
- [Derived] Giovannini-Chami L, Paquet A, Sanfiorenzo C, Pons N, Cazareth J, Magnone V, Lebrigand K, Chevalier B, Vallauri A, Julia V, Marquette CH, Marcet B, Leroy S, Barbry P. The "one airway, one disease" concept in light of Th2 inflammation. Eur Respir J. 2018 Oct 25;52(4):1800437. doi: 10.1183/13993003.00437-2018. Print 2018 Oct. PMID 30190271